CLINICAL TRIAL: NCT03449758
Title: Effect of Sarilumab on Patient-reported Outcomes in Patients With Moderately to Severely Active Rheumatoid Arthritis and With Inadequate Response or Intolerance to Current Conventional Synthetic DMARDs or Tumor Necrosis Factor Inhibitors
Brief Title: Effect of Sarilumab on Patient-reported Outcomes in Patients With Active Rheumatoid Arthritis
Acronym: SariPRO
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SARILL08755; U1111-1197-7699 (Other: UTN); 2017-002951-27 (EudraCT Number)
Record Dates: First submitted 2018-02-08; First posted 2018-02-28 (Actual); Results first posted 2020-08-10 (Actual); Last update posted 2022-04-28 (Actual); Status verified 2022-03

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — sarilumab; Azathioprine; Chloroquine; Hydroxychloroquine; Leflunomide; Methotrexate; Sulfasalazine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Sarilumab (Experimental): Sarilumab 200 milligram (mg) subcutaneous (SC) injection every 2 weeks (q2w) from Day 1 of Week 0 up to Week 24 as monotherapy and/or in combination with methotrexate (MTX) or other csDMARD during the randomized 6-month (24 weeks) core treatment period. Participants completing 24 weeks period entered in a long-term extension treatment period and received sarilumab 200 mg q2w from Week 25 until the commercial availability of sarilumab in the country or maximum of up to Week 39.7.
  Interventions: Drug: SARILUMAB; Drug: Azathioprine; Drug: Chloroquine; Drug: Hydroxychloroquine; Drug: Leflunomide; Drug: Methotrexate; Drug: Sulfasalazine

INTERVENTIONS:
Drug: SARILUMAB — Pharmaceutical form:Solution for injection in pre-filled syringe Route of administration: Subcutaneous
  Other Names: SAR153191 (REGN88); Kevzara®
Drug: Azathioprine — Pharmaceutical form:Tablet Route of administration: Oral
Drug: Chloroquine — Pharmaceutical form:Tablet Route of administration: Oral
Drug: Hydroxychloroquine — Pharmaceutical form:Tablet Route of administration: Oral
Drug: Leflunomide — Pharmaceutical form:Tablet Route of administration: Oral
Drug: Methotrexate — Pharmaceutical form:Solution for injection Route of administration: Subcutaneous / Intramuscular
Drug: Sulfasalazine — Pharmaceutical form:Tablet Route of administration: Oral

SUMMARY:
Primary Objective:

To assess the effect of sarilumab in combination with conventional synthetic Disease-Modifying Anti-Rheumatic Drug (csDMARD) and/or monotherapy on participant-reported impact of disease, using the rheumatoid arthritis impact of disease (RAID) questionnaire, in participants with moderately to severely active rheumatoid arthritis (RA) and inadequate response or intolerance to current csDMARD or tumor necrosis factor (TNF) inhibitors.

Secondary Objectives:

* To assess the change of the RAID score from baseline (to Week 4, Week 12, and Week 24) in participants with moderately to severely active RA and inadequate response or intolerance to current csDMARD or TNF inhibitors, treated with sarilumab in combination with csDMARD and/or monotherapy.
* To assess the effect of sarilumab in combination with csDMARD and/or monotherapy on other participant-reported outcomes (global assessment of disease activity, disability, morning stiffness, fatigue, anxiety/depression, mood disorders, and physical activities) in participants with moderately to severely active RA and inadequate response or intolerance to current csDMARD or TNF inhibitors.
* To assess the efficacy of sarilumab in combination with csDMARD and/or monotherapy using disease activity score-28 for RA with erythrocyte sedimentation rate (DAS28-ESR) and clinical disease activity index in participants with moderately to severely active RA and inadequate response or intolerance to current csDMARD or TNF inhibitors.
* To assess the safety of sarilumab in combination with csDMARD and/or monotherapy in participants with moderately to severely active RA and inadequate response or intolerance to current csDMARD or TNF inhibitors.

DETAILED DESCRIPTION:
The study duration per participant was approximately 32 weeks, with up to 4-week screening, 24 weeks treatment period, and 2-4 weeks post-treatment observations.

ELIGIBILITY:
Inclusion criteria :

* Participants with moderately to severely active RA to European League against Rheumatology (EULAR)/American College of Rheumatology (ACR) Criteria.
* Participants with moderate to severe disease activity defined as a DAS28-ESR greater than (>) 3.2 at Screening.
* Participants with inadequate response within at least the last 3 months or intolerance to current csDMARD or to at least one anti-TNF therapy (as defined by the investigator).
* Oral corticosteroids (less than or equal to [<=] 15 mg/day prednisone or equivalent) and nonsteroidal anti-inflammatory drugs or cyclooxygenase-2 (up to the maximum recommended dose) were allowed if taken at a stable dose for at least 4 weeks prior to Baseline.
* Permitted csDMARDs were allowed if taken at a stable dose for at least 4 weeks prior to Baseline.
* Participants abled and given written informed consent and complied with the requirements of the study protocol.

Exclusion criteria:

* Less than (<) 18 years of age.
* Participant unable to understand and write adequately to complete the study participant related outcome assessments.
* Exposure to sarilumab at any time prior to Baseline visit.
* Use of intra-articular or parenteral corticosteroids within 4 weeks prior to Baseline.
* Treatment with any investigational agent within the 4 weeks of Screening.
* Last RA treatment prior to inclusion with any anti-Janus kinase (JAK) or biologic DMARD other than anti-TNF.
* Participants treated with anti-TNF (i.e. adalimumab, infliximab, certolizumab, golimumab, etanercept) before the screening period, which are maintained within the 4 weeks before the inclusion (i.e. the first injection of sarilumab).
* Rheumatic autoimmune disease other than RA or prior history or current inflammatory joint disease other than RA.
* Evidence of active malignant disease, malignancies diagnosed within the previous 10 years (except basal and squamous cell carcinoma of the skin or carcinoma in situ of the cervix uteri previously excised and cured).
* Participant who was institutionalized due to regulatory or legal order or participant who was mentally disabled or educationally disadvantaged.
* Pregnant or breastfeeding woman.
* Women of childbearing potential not protected by highly-effective contraceptive method(s) of birth control (as defined in the informed consent form and/or in a local protocol addendum/amendment) over the study period and for at least 3 months following the last dose of sarilumab, and/or who are unwilling or unable to be tested for pregnancy.
* History of severe allergic or anaphylactic reactions to human, humanized, or murine monoclonal antibodies (or to any of the excipients associated to sarilumab).
* Immunization with a live/attenuated vaccine within 4 weeks prior to Baseline.
* Stage III or IV cardiac failure according to the New York Heart Association classification.
* History of previous gastrointestinal perforation or diverticulitis.
* Known active current/ recurrent infections (including but not limited to active tuberculosis [TB] or history of incompletely treated TB and atypical mycobacterial disease, hepatitis B and C, and herpes zoster). NOTE: in case of latent TB infection the participant might be included if a subsequent appropriate anti TB treatment is initiated since at least 3 weeks.
* Positive hepatitis B surface antigen, and/or positive total hepatitis B core antibody, and/or positive hepatitis C antibody at the Screening visit.
* Evidence of serious uncontrolled concomitant disease, including severe uncontrolled hypercholesterolemia or hypertriglyceridemia.
* Participants with any of the following laboratory abnormalities at the Screening or Baseline visit:

  * Hemoglobin <8.5 grams per deciliter.
  * White blood cells <3000/cubic millimeter (mm^3).
  * Absolute neutrophil count <2000/mm^3
  * Absolute lymphocyte count <500/mm^3
  * Platelet count <150 000 cells/mm^3
  * Creatinine clearance <30 milliliter per minute.
  * Aspartate aminotransaminase or Alanine aminotransaminase >1.5 x upper limit of normal (ULN).
  * Bilirubin (total) >ULN, unless Gilbert's disease has been determined by genetic testing and has been documented
  * Total fasting cholesterol >3.50 gram per liter (g/L) [9.1 millimoles per liter {mmol/L}]) or triglycerides >5.00 g/L [5.6 mmol/L]).

The above information was not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2018-03-05 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (33):
- France (33):
  - Investigational Site Number 250007, Argenteuil
  - Investigational Site Number 250006, Besançon
  - Investigational Site Number 250027, Bobigny
  - Investigational Site Number 250016, Bordeaux
  - Investigational Site Number 250014, Caen
  - Investigational Site Number 250032, Cahors
  - Investigational Site Number 250019, Cannes
  - Investigational Site Number 250013, Cholet
  - Investigational Site Number 250002, Clermont-Ferrand
  - Investigational Site Number 250009, Échirolles
  - Investigational Site Number 250005, La Roche-sur-Yon
  - Investigational Site Number 250024, Le Mans
  - Investigational Site Number 250004, Lille
  - Investigational Site Number 250012, Limoges
  - Investigational Site Number 250021, Lyon
  - Investigational Site Number 250018, Montivilliers
  - Investigational Site Number 250029, Montpellier
  - Investigational Site Number 250025, Nantes
  - Investigational Site Number 250026, Nice
  - Investigational Site Number 250010, Paris
  - Investigational Site Number 250011, Paris
  - Investigational Site Number 250015, Paris
  - Investigational Site Number 250028, Paris
  - Investigational Site Number 250020, Paris
  - Investigational Site Number 250033, Paris
  - Investigational Site Number 250031, Poitiers
  - Investigational Site Number 250023, Pontoise
  - Investigational Site Number 250017, Rennes
  - Investigational Site Number 250008, Rouen
  - Investigational Site Number 250001, Saint-Etienne
  - Investigational Site Number 250034, Strasbourg
  - Investigational Site Number 250022, Toulouse
  - Investigational Site Number 250003, Tours

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 31 active centers in France. A total of 104 participants were screened between 05 March 2018 to 27 December 2018, of which 20 were screen failures. Screen failures were mainly due to inclusion criteria not met.
Pre-assignment Details: A total of 84 participants were enrolled and received treatment.
Groups:
- Sarilumab: Sarilumab 200 mg subcutaneous (SC) injection every 2 weeks (q2w) from Day 1 of Week 0 up to Week 24 as monotherapy and/or in combination with methotrexate (MTX) or other conventional synthetic Disease-Modifying Antirheumatic Drugs (csDMARD) during the randomized 6-months (24 weeks) core treatment period. Participants completing 24 weeks period entered in a long-term extension treatment period and received sarilumab 200 mg q2w from Week 25 until the commercial availability of sarilumab in the country or maximum of up to Week 39.7.
Period: Overall Study
Arm/Group | Sarilumab
Started (Enrolled and treated.) | 84
Completed | 65
Not Completed | 19
Not completed — Major protocol deviation | 1
Not completed — Treatment inefficacy | 5
Not completed — Adverse Event | 9
Not completed — Consent withdrawal | 1
Not completed — Other unspecified reason | 3

BASELINE CHARACTERISTICS:
Population: Analysis was performed on intent-to-treat (ITT) population which included participants who met all the eligibility criteria and received study treatment at least once.
Groups:
- Sarilumab: Sarilumab 200 mg SC injection q2w from Day 1 of Week 0 up to Week 24 as monotherapy and/or in combination with MTX or other csDMARD during the randomized 6-month (24 weeks) core treatment period. Participants completing 24 weeks period entered in a long-term extension treatment period and received sarilumab 200 mg q2w from Week 25 until the commercial availability of sarilumab in the country or maximum of up to Week 39.7.
Arm/Group | Sarilumab
Number analyzed (Participants) | 84
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.1 (12.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 63
  Male | 21
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Rheumatoid Arthritis Impact of Disease (RAID) - Baseline Total Score [Mean (Standard Deviation); unit: score on a scale] — RAID is a participant-reported outcome measure used to evaluate impact of rheumatoid arthritis (RA) on participant's quality of life which comprised 7 domains: pain, function, fatigue, physical and psychological well-being, sleep disturbance, and coping. Each domain was a single question scored on 0 to 10 continuous numerical rating scale (NRS). Values for each of these domains were weighed by participant assessment of relative importance and combined in single value. Total RAID score range was 0 (not affected, very good) to 10 (most affected), where higher value indicated worse status.
  score on a scale | 5.8 (1.9)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Rheumatoid Arthritis Impact of Disease Total Score at Week 24
Description: RAID was a participant reported outcome measure used to evaluate the impact of RA on participant's quality of life which comprised 7 domains: • pain, • function, • fatigue, • physical and psychological well-being, • sleep disturbance, and • coping. Each domain was a single question scored on a 0 to 10 continuous NRS. The values for each of these domains were weighed by participant assessment of relative importance and combined in a single value. Total RAID score range was 0 (not affected, very good) to 10 (most affected), where higher value indicated worse status.
Time Frame: Baseline, Week 24
Population: Analysis was performed on ITT population. Here, 'overall number of participants analyzed' = participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Sarilumab: Sarilumab 200 mg SC injection q2w from Day 1 of Week 0 up to Week 24 as monotherapy and/or in combination with MTX or other csDMARD during the randomized 6-months (24 weeks) core treatment period. Participants completing 24 weeks period entered in a long-term extension treatment period and received sarilumab 200 mg q2w from Week 25 until the commercial availability of sarilumab in the country or maximum of up to Week 39.7.
Arm/Group | Sarilumab
Number analyzed (Participants) | 62
score on a scale | -2.4 (2.3)

2. Secondary Outcome: Rheumatoid Arthritis Impact of Disease Total Score at Baseline, Weeks 4, 12 and 24
Description: RAID was a participant reported outcome measure used to evaluate the impact of RA on participant's quality of life which comprised 7 domains: • pain, • function, • fatigue, • physical and psychological well-being, • sleep disturbances, and • coping. Each domain was a single question scored on a 0 to 10 continuous NRS. The values for each of these domains were weighed by participant assessment of relative importance and combined in a single value. Total RAID score range was 0 (not affected, very good) to 10 (most affected), where higher value indicated worse status.
Time Frame: Baseline, Weeks 4, 12 and 24
Population: Analysis was performed on ITT population. Here, 'number analyzed' = participants with available data for each specified category.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sarilumab
Number analyzed (Participants) | 84
score on a scale
  Week 4: number analyzed (Participants) | 82
  Week 4 | 4.6 (2.1)
  Week 12: number analyzed (Participants) | 70
  Week 12 | 3.9 (2.3)
  Week 24: number analyzed (Participants) | 64
  Week 24 | 3.3 (2.5)

3. Secondary Outcome: Change From Baseline in Rheumatoid Arthritis Impact of Disease Total Score at Weeks 4 and 12
Description: RAID was a participant reported outcome measure used to evaluate the impact of RA on participant's quality of life which comprised 7 domains: • pain, • function, • fatigue, • physical and psychological wellbeing, • sleep disturbance, and • coping. Each domain was a single question scored on a 0 to 10 continuous NRS. The values for each of these domains were weighed by participant assessment of relative importance and combined in a single value. Total RAID score range was 0 (not affected, very good) to 10 (most affected), where higher value indicated worse status.
Time Frame: Baseline, Weeks 4 and 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sarilumab
Number analyzed (Participants) | 84
score on a scale
  Week 4: number analyzed (Participants) | 80
  Week 4 | -1.2 (1.6)
  Week 12: number analyzed (Participants) | 68
  Week 12 | -1.8 (2.2)

4. Secondary Outcome: Hospital Anxiety and Depression Scale (HADS): Anxiety (HADS-A) and Depression (HADS-D) Subscale Scores at Baseline, Weeks 4, 12, and 24
Description: HADS questionnaire measures the presence and severity of anxiety and depression in both hospital and community settings. The questionnaire comprised of 14 items divided into 2 subscales: 7 items for anxiety subscale (HADS-A) and 7 items for depression subscale (HADS-D). Each item was scored on a 0 to 3 rating scale. The anxiety and depression subscales each ranged from 0 to 21 (0-7: normal, 8-10: borderline abnormal and 11-21: abnormal), where higher scores indicated greater severity of anxiety/depression. The subscales were independent for each result of depression and anxiety.
Time Frame: Baseline, Weeks 4, 12 and 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Sarilumab: Sarilumab 200 mg SC injection q2w from Day 1 of Week 0 up to Week 24 as monotherapy and/or in combination with MTX or other csDMARD during the randomized 6-months core treatment period. Participants who completed the 24 weeks period had an option to continue in a long-term extension treatment period and received sarilumab 200 mg q2w until the commercial availability of sarilumab in the country or maximum of 39.7 weeks.
Arm/Group | Sarilumab
Number analyzed (Participants) | 84
score on a scale
  HADS-A: Baseline: number analyzed (Participants) | 80
  HADS-A: Baseline | 8.1 (4.3)
  HADS-A: Week 4: number analyzed (Participants) | 76
  HADS-A: Week 4 | 7.2 (4.3)
  HADS-A: Week 12: number analyzed (Participants) | 68
  HADS-A: Week 12 | 6.1 (3.7)
  HADS-A: Week 24: number analyzed (Participants) | 61
  HADS-A: Week 24 | 6.6 (3.9)
  HADS-D: Baseline: number analyzed (Participants) | 82
  HADS-D: Baseline | 7.0 (3.9)
  HADS-D: Week 4: number analyzed (Participants) | 79
  HADS-D: Week 4 | 6.6 (4.0)
  HADS-D: Week 12: number analyzed (Participants) | 70
  HADS-D: Week 12 | 5.7 (4.1)
  HADS-D: Week 24: number analyzed (Participants) | 61
  HADS-D: Week 24 | 5.5 (4.1)

5. Secondary Outcome: Change From Baseline in Hospital Anxiety and Depression Scale: Anxiety (HADS-A) and Depression (HADS-D) Subscale Scores at Weeks 4, 12 and 24
Description: as for outcome 4
Time Frame: Baseline, Weeks 4, 12 and 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sarilumab
Number analyzed (Participants) | 84
score on a scale
  HADS-A: Week 4: number analyzed (Participants) | 72
  HADS-A: Week 4 | -1.0 (2.4)
  HADS-A: Week 12: number analyzed (Participants) | 65
  HADS-A: Week 12 | -2.1 (3.3)
  HADS-A: Week 24: number analyzed (Participants) | 57
  HADS-A: Week 24 | -1.9 (3.2)
  HADS-D: Week 4: number analyzed (Participants) | 77
  HADS-D: Week 4 | -0.4 (2.5)
  HADS-D: Week 12: number analyzed (Participants) | 69
  HADS-D: Week 12 | -1.2 (4.1)
  HADS-D: Week 24: number analyzed (Participants) | 59
  HADS-D: Week 24 | -1.7 (3.7)

6. Secondary Outcome: Multidimensional Assessment of Thymic States (MAThyS) Scale Total Score at Baseline, Weeks 4, 12 and 24
Description: MAThyS was a multi-dimensional self-administered questionnaire comprised of five dimensions (emotional reactivity, cognition speed, psychomotor function, motivation and sensory perception) divided into 20 items relating to individual states as perceived by participants for the preceding week (at each specified Week). Each item was measured on a visual analog scale (VAS; in centimeters [cm]) ranged from 0 (inhibition of the state evaluated by the item) to 10 (excitation for the evaluated state). Total MAThyS score was sum of the 20 items and that might vary from score range 0 to 200 with lower scores indicated general inhibition and higher scores indicated general excitation.
Time Frame: Baseline, Weeks 4, 12 and 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Sarilumab
Number analyzed (Participants) | 84
cm
  Baseline: number analyzed (Participants) | 80
  Baseline | 88.4 (21.1)
  Week 4: number analyzed (Participants) | 79
  Week 4 | 89.6 (20.3)
  Week 12: number analyzed (Participants) | 72
  Week 12 | 94.8 (13.6)
  Week 24: number analyzed (Participants) | 66
  Week 24 | 90.9 (22.3)

7. Secondary Outcome: Change From Baseline in Multidimensional Assessment of Thymic States Scale Total Score at Weeks 4, 12 and 24
Description: MAThyS was a multi-dimensional self-administered questionnaire comprised of five dimensions (emotional reactivity, cognition speed, psychomotor function, motivation and sensory perception) divided into 20 items relating to individual states as perceived by participants for the preceding week (at each specified Week). Each item was measured on a VAS (in cm) ranging from 0 (inhibition of the state evaluated by the item) to 10 (excitation for the evaluated state). Total MAThyS score was sum of the 20 items and that might vary from score range 0 to 200 with lower scores indicated general inhibition and higher scores indicated general excitation.
Time Frame: Baseline, Weeks 4, 12 and 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Sarilumab
Number analyzed (Participants) | 84
cm
  Week 4: number analyzed (Participants) | 76
  Week 4 | -0.2 (24.2)
  Week 12: number analyzed (Participants) | 70
  Week 12 | 2.9 (17.7)
  Week 24: number analyzed (Participants) | 63
  Week 24 | -1.1 (23.4)

8. Secondary Outcome: Functional Assessment of Chronic Illness Therapy - Fatigue (FACIT-F) Total Scores at Baseline, Weeks 4, 12 and 24
Description: FACIT-F was a 13-item questionnaire that assess fatigue in participants under chronic illness therapy. Participants scored each item on a 5-point Likert scale ranged from 0 to 4 (0 = not at all; 1 = a little bit; 2 = somewhat; 3 = quite a bit; 4 = very much). The scores of each item were reversed during score calculations, so that higher score values indicated more favorable conditions. Total score was the sum of score from each item and resulted in a score range from 0 to 52, with higher score indicated better participant health status (lower level of fatigue).
Time Frame: Baseline, Weeks 4, 12 and 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sarilumab
Number analyzed (Participants) | 84
score on a scale
  Baseline: number analyzed (Participants) | 82
  Baseline | 25.5 (10.3)
  Week 4: number analyzed (Participants) | 83
  Week 4 | 21.0 (10.5)
  Week 12: number analyzed (Participants) | 74
  Week 12 | 18.8 (9.7)
  Week 24: number analyzed (Participants) | 66
  Week 24 | 17.9 (11.4)

9. Secondary Outcome: Change From Baseline in Functional Assessment of Chronic Illness Therapy - Fatigue Total Scores at Weeks 4, 12 and 24
Description: as for outcome 8
Time Frame: Baseline, Weeks 4, 12 and 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sarilumab
Number analyzed (Participants) | 84
score on a scale
  Week 4: number analyzed (Participants) | 81
  Week 4 | -4.8 (8.0)
  Week 12: number analyzed (Participants) | 72
  Week 12 | -6.4 (9.1)
  Week 24: number analyzed (Participants) | 64
  Week 24 | -7.6 (10.8)

10. Secondary Outcome: Stanford Health Assessment Questionnaire Disability Index (HAQ-DI) Total Score at Baseline, Weeks 4, 12 and 24
Description: HAQ-DI was a participant-oriented questionnaire developed specifically to assess the extent of a RA participant's functional ability. It consisted of at least 2 or 3 questions per category, participant reported assessment of ability to perform tasks in 8 categories of daily living activities: dress/groom; arise; eat; walk; reach; grip; hygiene; and common activities over past week (at each specified visit) rated on a 4-point scale where 0 = no difficulty; 1 = some difficulty; 2 = much difficulty; 3 = unable to do. Overall score was computed as the sum of category scores and divided by the number of categories answered, and ranged from 0 to 3, where 0 = no disability and 3 = completely disabled, higher score indicated more disability.
Time Frame: Baseline, Weeks 4, 12 and 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sarilumab
Number analyzed (Participants) | 84
score on a scale
  Baseline: number analyzed (Participants) | 82
  Baseline | 1.3 (0.8)
  Week 4: number analyzed (Participants) | 81
  Week 4 | 1.1 (0.7)
  Week 12: number analyzed (Participants) | 74
  Week 12 | 0.8 (0.7)
  Week 24: number analyzed (Participants) | 67
  Week 24 | 0.8 (0.8)

11. Secondary Outcome: Change From Baseline in Stanford Health Assessment Questionnaire Disability Index Total Score at Weeks 4, 12 and 24
Description: as for outcome 10
Time Frame: Baseline, Weeks 4, 12 and 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sarilumab
Number analyzed (Participants) | 84
score on a scale
  Week 4: number analyzed (Participants) | 79
  Week 4 | -0.2 (0.5)
  Week 12: number analyzed (Participants) | 72
  Week 12 | -0.4 (0.6)
  Week 24: number analyzed (Participants) | 65
  Week 24 | -0.5 (0.8)

12. Secondary Outcome: Duration of Morning Stiffness at Baseline, Weeks 4, 12, and 24
Description: Duration of morning stiffness was defined as the time elapsed (in minutes) between the time of usual awakening (even if not in the morning) and the time the participant was able to resume normal activities without stiffness. At each specified time point, duration of morning stiffness was reported by the participant during the visit.
Time Frame: Baseline, Weeks 4, 12 and 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Sarilumab
Number analyzed (Participants) | 84
minutes
  Baseline: number analyzed (Participants) | 79
  Baseline | 72.3 (75.0)
  Week 4: number analyzed (Participants) | 78
  Week 4 | 34.7 (43.9)
  Week 12: number analyzed (Participants) | 76
  Week 12 | 28.9 (47.2)
  Week 24: number analyzed (Participants) | 68
  Week 24 | 21.3 (37.5)

13. Secondary Outcome: Change From Baseline in Duration of Morning Stiffness at Weeks 4, 12, and 24
Description: as for outcome 12
Time Frame: Baseline, Weeks 4, 12 and 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Sarilumab
Number analyzed (Participants) | 84
minutes
  Week 4: number analyzed (Participants) | 74
  Week 4 | -39.9 (67.9)
  Week 12: number analyzed (Participants) | 71
  Week 12 | -47.9 (76.8)
  Week 24: number analyzed (Participants) | 63
  Week 24 | -52.8 (72.3)

14. Secondary Outcome: International Physical Activity Questionnaire (IPAQ) Total Score at Baseline, Weeks 4, 12 and 24
Description: IPAQ was a 27-item self-reported questionnaire designed to measure physical activity of participant. The score was reported in metabolic equivalent (MET)-minutes per week. MET minutes represented the amount of energy expended to carry out physical activity. For IPAQ total score, the minimum value is zero and there is no maximum. Higher scores mean better levels of physical activity.
Time Frame: Baseline, Weeks 4, 12 and 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: MET minutes per week
Arm/Group | Sarilumab
Number analyzed (Participants) | 84
MET minutes per week
  Baseline: number analyzed (Participants) | 52
  Baseline | 1759.9 (1185.0)
  Week 4: number analyzed (Participants) | 57
  Week 4 | 1881.1 (1203.9)
  Week 12: number analyzed (Participants) | 50
  Week 12 | 2061.0 (1266.9)
  Week 24: number analyzed (Participants) | 47
  Week 24 | 2089.5 (1476.4)

15. Secondary Outcome: Change From Baseline in International Physical Activity Questionnaire Total Score at Weeks 4, 12 and 24
Description: IPAQ was a 27-item self-reported questionnaire designed to measure physical activity of participant. The score was reported in MET minutes per week. MET minutes represented the amount of energy expended to carry out physical activity. For IPAQ total score, the minimum value is zero and there is no maximum. Higher scores mean better levels of physical activity.
Time Frame: Baseline, Weeks 4, 12 and 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: MET minutes per week
Arm/Group | Sarilumab
Number analyzed (Participants) | 84
MET minutes per week
  Week 4: number analyzed (Participants) | 42
  Week 4 | 175.6 (1177.7)
  Week 12: number analyzed (Participants) | 38
  Week 12 | 533.4 (1509.7)
  Week 24: number analyzed (Participants) | 33
  Week 24 | 382.0 (1719.8)

16. Secondary Outcome: Patient Global Assessment (PtGA) of Disease Activity Score by Visual Analog Scale (VAS) at Baseline, Weeks 4, 12 and 24
Description: PtGA of disease activity was measured using a 100 millimeters (mm) horizontal VAS ranged from 0=no pain to 100=maximum pain imaginable, where higher score indicated more disease activity.
Time Frame: Baseline, Weeks 4, 12 and 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Sarilumab
Number analyzed (Participants) | 84
mm
  Baseline | 61.1 (22.4)
  Week 4: number analyzed (Participants) | 83
  Week 4 | 44.1 (25.6)
  Week 12: number analyzed (Participants) | 78
  Week 12 | 36.6 (26.7)
  Week 24: number analyzed (Participants) | 69
  Week 24 | 34.6 (25.6)

17. Secondary Outcome: Change From Baseline in Patient Global Assessment of Disease Activity Score by Visual Analog Scale at Weeks 4, 12, and 24
Description: PtGA of disease activity was measured using a 100 mm horizontal VAS ranged from 0=no pain to 100=maximum pain imaginable, where higher score indicated more disease activity.
Time Frame: Baseline, Weeks 4, 12 and 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Sarilumab
Number analyzed (Participants) | 84
mm
  Week 4: number analyzed (Participants) | 83
  Week 4 | -17.2 (24.2)
  Week 12: number analyzed (Participants) | 78
  Week 12 | -24.3 (31.8)
  Week 24: number analyzed (Participants) | 69
  Week 24 | -26.7 (29.6)

18. Secondary Outcome: Erythrocyte Sedimentation Rate (ESR) at Baseline, Weeks 4, 12, and 24
Description: ESR was a laboratory test to provide non-specific measure of inflammation in the body. The test assessed the rate at which red blood cells fell in a test tube and was measured in millimeter per hour (mm/h).
Time Frame: Baseline, Weeks 4, 12 and 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mm/h
Arm/Group | Sarilumab
Number analyzed (Participants) | 84
mm/h
  Baseline: number analyzed (Participants) | 82
  Baseline | 28.8 (23.4)
  Week 4: number analyzed (Participants) | 83
  Week 4 | 10.5 (15.5)
  Week 12: number analyzed (Participants) | 78
  Week 12 | 9.2 (15.3)
  Week 24: number analyzed (Participants) | 67
  Week 24 | 8.4 (11.3)

19. Secondary Outcome: Change From Baseline in Erythrocyte Sedimentation Rate at Weeks 4, 12, and 24
Description: ESR was a laboratory test to provide non-specific measure of inflammation in the body. The test assessed the rate at which red blood cells fell in a test tube and was measured in mm/h.
Time Frame: Baseline, Weeks 4, 12 and 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mm/h
Arm/Group | Sarilumab
Number analyzed (Participants) | 84
mm/h
  Week 4: number analyzed (Participants) | 81
  Week 4 | -18.1 (21.1)
  Week 12: number analyzed (Participants) | 77
  Week 12 | -19.5 (25.1)
  Week 24: number analyzed (Participants) | 66
  Week 24 | -22.0 (23.2)

20. Secondary Outcome: Disease Activity Score-28 for Rheumatoid Arthritis With Erythrocyte Sedimentation Rate (DAS28-ESR) at Baseline, Weeks 4, 12, and 24
Description: DAS28-ESR was a composite score that included 4 variables: tender joint count (TJC) (based on 28 joints); swollen joint count (SJC) (based on 28 joints); participant's global assessment of health activity using 100 mm VAS: range 0 (no pain) to 100 (maximum pain imaginable); marker of inflammation assessed by ESR in mm/h. DAS28-ESR total score ranged from 0-10, higher score indicated more disease activity. The DAS28-ESR score provided a number indicating the current disease activity of the RA. A DAS28-ESR score above 5.1 indicated high disease activity, DAS28-ESR score less than or equal to (<=) 3.2 indicated low disease activity (LDA), greater than (>) 3.2 to <=5.1 implied moderate disease activity and DAS28-ESR score below 2.6 indicated disease remission.
Time Frame: Baseline, Weeks 4, 12 and 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sarilumab
Number analyzed (Participants) | 84
score on a scale
  Baseline: number analyzed (Participants) | 82
  Baseline | 5.0 (1.2)
  Week 4: number analyzed (Participants) | 83
  Week 4 | 3.1 (1.5)
  Week 12: number analyzed (Participants) | 78
  Week 12 | 2.6 (1.5)
  Week 24: number analyzed (Participants) | 67
  Week 24 | 2.3 (1.4)

21. Secondary Outcome: Change From Baseline in Disease Activity Score-28 for Rheumatoid Arthritis With Erythrocyte Sedimentation Rate at Weeks 4, 12, and 24
Description: DAS28-ESR was a composite score that included 4 variables: TJC (based on 28 joints); SJC (based on 28 joints); participant's global assessment of health activity using 100 mm VAS: range 0 (no pain) to 100 (maximum pain imaginable); marker of inflammation assessed by ESR in mm/h. DAS28-ESR total score ranged from 0-10, higher score indicated more disease activity. The DAS28-ESR score provided a number indicating the current disease activity of the RA. A DAS28-ESR score above 5.1 indicated high disease activity, DAS28-ESR score <= 3.2 indicated LDA, > 3.2 to <=5.1 implied moderate disease activity and DAS28-ESR score below 2.6 indicated disease remission.
Time Frame: Baseline, Weeks 4, 12 and 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sarilumab
Number analyzed (Participants) | 84
score on a scale
  Week 4: number analyzed (Participants) | 81
  Week 4 | -1.8 (1.1)
  Week 12: number analyzed (Participants) | 77
  Week 12 | -2.3 (1.6)
  Week 24: number analyzed (Participants) | 66
  Week 24 | -2.7 (1.5)

22. Secondary Outcome: Clinical Disease Activity Index (CDAI) Total Score at Baseline, Weeks 4, 12, and 24
Description: CDAI was a composite index constructed to measure clinical remission in RA that does not include a laboratory test, and is a numerical summation of 4 components: SJC (28 joints), TJC (28 joints), participant's global disease activity (in cm), and physician's global assessment of disease (in cm). CDAI total score ranges from 0 to 76 with a lower score indicating less disease activity. A CDAI score of <=2.8 represents clinical remission and a score of <=10.0 represents LDA.
Time Frame: Baseline, Weeks 4, 12 and 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sarilumab
Number analyzed (Participants) | 84
score on a scale
  Baseline: number analyzed (Participants) | 82
  Baseline | 22.5 (11.2)
  Week 4: number analyzed (Participants) | 83
  Week 4 | 12.6 (9.8)
  Week 12: number analyzed (Participants) | 78
  Week 12 | 9.9 (10.4)
  Week 24: number analyzed (Participants) | 67
  Week 24 | 8.1 (7.8)

23. Secondary Outcome: Change From Baseline in Clinical Disease Activity Index Total Score at Weeks 4, 12, and 24
Description: as for outcome 22
Time Frame: Baseline, Weeks 4, 12 and 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sarilumab
Number analyzed (Participants) | 84
score on a scale
  Week 4: number analyzed (Participants) | 81
  Week 4 | -9.8 (8.1)
  Week 12: number analyzed (Participants) | 77
  Week 12 | -12.2 (13.2)
  Week 24: number analyzed (Participants) | 66
  Week 24 | -14.6 (12.6)

24. Secondary Outcome: Number of Swollen Joints at Baseline, Weeks 4, 12, and 24
Description: Number of joints with swelling are reported. Joints which were assessed included 28 joints (which included shoulders, elbows, wrists, knees and 2 joints in each finger and thumb).
Time Frame: Baseline, Weeks 4, 12 and 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: joints
Arm/Group | Sarilumab
Number analyzed (Participants) | 84
joints
  Baseline: number analyzed (Participants) | 83
  Baseline | 6.3 (5.1)
  Week 4: number analyzed (Participants) | 83
  Week 4 | 2.5 (3.2)
  Week 12: number analyzed (Participants) | 79
  Week 12 | 1.9 (3.6)
  Week 24: number analyzed (Participants) | 70
  Week 24 | 1.6 (2.8)

25. Secondary Outcome: Change From Baseline in Number of Swelling Joints at Weeks 4, 12, and 24
Description: as for outcome 24
Time Frame: Baseline, Weeks 4, 12 and 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: joints
Arm/Group | Sarilumab
Number analyzed (Participants) | 84
joints
  Week 4: number analyzed (Participants) | 82
  Week 4 | -3.9 (4.3)
  Week 12: number analyzed (Participants) | 78
  Week 12 | -4.1 (5.1)
  Week 24: number analyzed (Participants) | 69
  Week 24 | -4.7 (5.2)

26. Secondary Outcome: Number of Tender Joints at Baseline, Weeks 4, 12, and 24
Description: Number of joints with tenderness are reported. Joints which were assessed included 28 joints (which included shoulders, elbows, wrists, knees and 2 joints in each finger and thumb).
Time Frame: Baseline, Weeks 4, 12 and 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: joints
Arm/Group | Sarilumab
Number analyzed (Participants) | 84
joints
  Baseline: number analyzed (Participants) | 83
  Baseline | 7.3 (5.8)
  Week 4: number analyzed (Participants) | 83
  Week 4 | 4.7 (5.4)
  Week 12: number analyzed (Participants) | 79
  Week 12 | 3.5 (5.2)
  Week 24: number analyzed (Participants) | 70
  Week 24 | 2.5 (4.1)

27. Secondary Outcome: Change From Baseline in Number of Tender Joints at Weeks 4, 12, and 24
Description: as for outcome 26
Time Frame: Baseline, Weeks 4, 12 and 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: joints
Arm/Group | Sarilumab
Number analyzed (Participants) | 84
joints
  Week 4: number analyzed (Participants) | 82
  Week 4 | -2.5 (4.5)
  Week 12: number analyzed (Participants) | 78
  Week 12 | -3.7 (6.5)
  Week 24: number analyzed (Participants) | 69
  Week 24 | -4.8 (6.4)

28. Secondary Outcome: Number of Participants Achieving Low Disease Activity (DAS28 ESR Score <=3.2) and Remission (DAS28 ESR Score <2.6) at Weeks 12, and 24
Description: DAS28-ESR was a composite score that included 4 variables: TJC (based on 28 joints); SJC (based on 28 joints); participant's global assessment of health activity using 100 mm VAS: range 0 (no pain) to 100 (maximum pain imaginable) marker of inflammation assessed by ESR in mm/h. DAS28-ESR total score ranged from 0-10, higher score indicated more disease activity. The DAS28-ESR score provided a number indicating the current disease activity of the RA. A DAS28-ESR score above 5.1 indicated high disease activity, DAS28-ESR score <= 3.2 indicated LDA, > 3.2 to <=5.1 implied moderate disease activity and DAS28-ESR score below 2.6 indicated disease remission.
Time Frame: Weeks 12 and 24
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Sarilumab
Number analyzed (Participants) | 84
Participants
  LDA: Week 12: number analyzed (Participants) | 78
  LDA: Week 12 | 12
  LDA: Week 24: number analyzed (Participants) | 67
  LDA: Week 24 | 4
  Remission: Week 12: number analyzed (Participants) | 78
  Remission: Week 12 | 40
  Remission: Week 24: number analyzed (Participants) | 67
  Remission: Week 24 | 45

29. Secondary Outcome: Number of Participants Achieving Clinical Disease Activity Index: Low Disease Activity (CDAI Score <=10.0) and Remission (CDAI Score <=2.8) Weeks 12, and 24
Description: CDAI was a composite index constructed to measure clinical remission in RA that does not included a laboratory test, and is a numerical summation of 4 components: SJC (28 joints), TJC (28 joints), participant's global disease activity (in cm), and physician's global assessment (in cm). Total score ranged from 0 to 76 with a lower score indicated less disease activity. A CDAI score of <=2.8 represents clinical remission and a score of <=10.0 represents LDA.
Time Frame: Weeks 12 and 24
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Sarilumab
Number analyzed (Participants) | 84
Participants
  LDA: Week 12: number analyzed (Participants) | 78
  LDA: Week 12 | 29
  LDA: Week 24: number analyzed (Participants) | 67
  LDA: Week 24 | 29
  Remission: Week 12: number analyzed (Participants) | 78
  Remission: Week 12 | 18
  Remission: Week 24: number analyzed (Participants) | 67
  Remission: Week 24 | 20

30. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Description: An adverse event (AE) was defined as any untoward medical occurrence in a participant who received study drug and did not necessarily had a causal relationship with the study treatment. SAE: Any untoward medical occurrence that resulted in any of the following outcomes: death, life-threatening, required initial or prolonged in-patient hospitalization, persistent or significant disability/incapacity, congenital anomaly/birth defect, or considered as medically important event. TEAEs were defined as AEs that occurred in the time from the first injection of study drug up to 39.7 weeks.
Time Frame: Baseline up to end of study (up to 39.7 weeks)
Population: Analysis was performed on safety population which included participants who signed the informed consent form and had exposed to at least one dose or part of a dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Sarilumab
Number analyzed (Participants) | 84
Participants
  SAE | 10
  TEAE | 76
  AE leading to death | 0

ADVERSE EVENTS:
Time Frame: All AEs were collected from the time of first injection of study drug up to 39.7 weeks regardless of seriousness or relationship to study drug.
Description: Reported AEs were TEAEs which were defined as AEs that occurred in the time from the first injection of study drug up to 39.7 weeks. Analysis was performed on safety population.
Groups:
- Sarilumab: Sarilumab 200 mg SC injection q2w from Day 1 of Week 0 up to Week 24 as monotherapy and/or in combination with MTX or other csDMARD during the randomized 6-months (24 weeks) core treatment period. Participants completing 24 weeks period entered in a long-term extension treatment period and received sarilumab 200 mg q2w from Week 25 until the commercial availability of sarilumab in the country or maximum of up to 39.7 weeks.
Arm/Group | Sarilumab
All-Cause Mortality (participants affected / at risk) | 0/84
Serious Adverse Events (participants affected / at risk) | 10/84
Other Adverse Events (participants affected / at risk) | 54/84
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sarilumab (N=84)
Neutropenia (Blood and lymphatic system disorders) | 1 (2)
Drug Hypersensitivity (Immune system disorders) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Diabetes Mellitus Inadequate Control (Metabolism and nutrition disorders) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Lumbar Spinal Stenosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Rheumatoid Arthritis (Musculoskeletal and connective tissue disorders) | 1 (2)
Polyneuropathy (Nervous system disorders) | 1 (1)
Interstitial Lung Disease (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Angioedema (Skin and subcutaneous tissue disorders) | 1 (2)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sarilumab (N=84)
Neutropenia (Blood and lymphatic system disorders) | 16 (19)
Diarrhoea (Gastrointestinal disorders) | 5 (5)
Nausea (Gastrointestinal disorders) | 10 (11)
Asthenia (General disorders) | 9 (10)
Fatigue (General disorders) | 9 (9)
Injection Site Erythema (General disorders) | 5 (7)
Injection Site Pruritus (General disorders) | 5 (6)
Bronchitis (Infections and infestations) | 10 (11)
Nasopharyngitis (Infections and infestations) | 9 (10)
Headache (Nervous system disorders) | 9 (10)
Pruritus (Skin and subcutaneous tissue disorders) | 6 (6)

LIMITATIONS AND CAVEATS:
Secondary efficacy analyses was planned to be performed on the Per-protocol population (PPS), only when PPS represented less than 90 percent of the ITT population.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor supports publication of clinical trial results but may request that investigators temporarily delay or alter publications in order to protect proprietary information. The Sponsor may also require that the results of multicenter studies be published only in their entirety and not as individual site data.

DOCUMENTS (2):
  • Study Protocol (2018-06-06): https://cdn.clinicaltrials.gov/large-docs/58/NCT03449758/Prot_000.pdf
  • Statistical Analysis Plan (2019-11-19): https://cdn.clinicaltrials.gov/large-docs/58/NCT03449758/SAP_001.pdf